CLINICAL TRIAL: NCT04392206
Title: A Phase I, Open Label Study of Allogeneic Adipose Derived Mesenchymal Stem Cells in Reducing Anastomotic Stenosis in Primary Arteriovenous Anastomoses
Brief Title: AMSC for Reducing Anastomotic Stenosis in Primary Arteriovenous Anastomoses
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Houssam Farres, M.D. (Other)
Responsible Party: Sponsor-Investigator, Houssam Farres, M.D., Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-007203
Record Dates: First submitted 2020-05-14; First posted 2020-05-18 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adipose Derived Mesenchymal Stem Cells (Experimental): Subjects diagnosed with End Stage Renal Disease (ESRD) and are currently on hemodialysis therapy with planned creation of a new upper extremity arteriovenous fistula will receive Adipose Derived Mesenchymal Stem Cells treatment.
  Interventions: Drug: Adipose Derived Mesenchymal Stem Cells

INTERVENTIONS:
Drug: Adipose Derived Mesenchymal Stem Cells — The dose will be specifically tailored to each subject's vascular anatomy determined by the surgeon through ultrasound measurements. Approximately 3-5 million cells in 5ml Ringer Lactate (RL) Solution
  Other Names: AMSC

SUMMARY:
Researchers are evaluating the safety of allogeneic Adipose Derived Mesenchymal Stem Cells (AMSC) use during hemodialysis arteriovenous fistula and arterial bypass creation and its efficacy on improving access maturation and primary anastomotic patency.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 and 85 years old
* Patient currently planned for creation of an upper extremity AV fistula with suitable anatomy
* Ability to communicate meaningfully with investigative staff, competence to give written informed consent, and ability to comply with entire study procedures
* Life expectancy of at least 24 months
* If female, must be post-menopausal or not able to have children. Post-menopausal/non-child bearing status must be clearly documented in the medical record. If documentation of post-menopausal/non-child bearing status is not available then a pregnancy test must be performed.

Exclusion Criteria:

* Malignancy or treatment for malignancy within the previous 6 months
* Immunodeficiency including AIDS / HIV or Active autoimmune disease
* Documented hypercoagulable state or history of 2 or more DVTs or other spontaneous intravascular thrombotic events
* Treatment with any investigational drug/ device within 60 days prior to study entry or Any other condition which in the judgment of the investigator would preclude adequate evaluation of the safety and efficacy of AMSCs and the AVF
* History of failed organ transplant on immunosuppression.
* Subjects with known active infection (infection which is being treated)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | 12 months
  Evaluate the safety of AMSC administration by assessing the number of participants to experience an adverse event as defined by inflammation, infection (local or systemic), aneurysm formation, clinically significant increase or decrease in blood flow or thrombosis formation as evaluated through physical exam and ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Houssam Farres, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No